CLINICAL TRIAL: NCT03251196
Title: TB Sequel: Pathogenesis and Risk Factors of Long-term Sequelae of Pulmonary TB Defining Individual Outcomes and Public Health Impact
Brief Title: TB Sequel: Pathogenesis and Risk Factors of Long-term Sequelae of Pulmonary TB
Acronym: TBSEQUEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Research Center Borstel (Other); University of Witwatersrand, South Africa (Other); Mbeya Medical Research Centre NIMR (Unknown); Ministry of Health Instituto Nacional de Saude (Unknown); Medical Research Council Unit, The Gambia (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: LMU-IMPH-TB Sequel-01
Record Dates: First submitted 2017-07-31; First posted 2017-08-16 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Tract Infections; Tuberculosis, Pulmonary
MeSH Terms: conditions — Respiratory Tract Infections; Tuberculosis, Pulmonary | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Collection Bloods, Urine and Sputum will be obtained from each patient at different time-points for analysis and storage. They will include, but are not limited to: native urine, native sputum, extracted DNA from positive liquid culture, sputum pellet and surpernatant and whole blood (PAXgene, plasma, serum, PBMC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention, and Observational Study — Observational Study
  Other Names: Observational Study

SUMMARY:
This is an observational cohort study. Pulmonary tuberculosis (TB) patients will be enrolled at the time of TB diagnosis and prospectively followed for at least two years after TB-treatment initiation with optional prolonged follow-up. Study visits will be performed in the study clinics or if necessary at the participant's home at pre-defined time points after TB treatment initiation. Clinical assessments, biological sample collections and collection of socio-economic data will be performed according to the pre-defined schedule of events.

DETAILED DESCRIPTION:
The African continent today is emblematic of TB as a global health emergency with little known about the long-term sequelae. It is likely that TB patients from resource-constrained settings, who usually present with more extensive disease, are left with greater lung impairment.

This project aims to advance the understanding of the clinical, microbiologic, and host immune factors affecting the long-term sequelae of pulmonary tuberculosis; to identify the most important factors that contribute to lung impairment, including the immunological response and genetic predisposition of the host and differences in the biology of the pathogen; to determine occurrence of reversible and irreversible costs and socioeconomic consequences for patients; and to facilitate novel interventions to restore and preserve overall health, well-being and financial protection in patients with TB.

The core of the current project is a prospective cohort of up to 1600 patients across four countries (Mozambique, Tanzania, South Africa and The Gambia), enrolled at the time of TB diagnosis, and followed up for at least 2 years. The overall goal of the cohort is to describe and analyse the basis of the long-term clinical consequences of pulmonary TB, with a particular focus on lung injury. The investigators will enroll patients during two years and follow each patient up for at least two years. The project also includes a number of sub-studies: Host-Immunology, Pathogen and Socio-Economic. General laboratory tests and TB specific tests, X-ray, physical examination and cardio-pulmonary assessment will be performed and the obtained clinical data will be recorded in study questionnaires. The investigators will collect and analyse biological specimens (blood, urine and sputum) longitudinally during the period of observation and after all specimens have been stored. In-depth analysis of the host immune response, focusing on potential mechanisms of lung damage, including oxidative injury, proteolytic matrix degradation, and neutrophil-mediated damage, neutrophil-macrophage ratios and markers; and molecular analysis of mycobacterial dynamics and markers in relation to pulmonary and microbiological treatment outcomes, including success, failure, relapse, reinfection and death will be carried out. Socio-economic data, including patient costs, will be collected at the time of TB diagnosis, during treatment, at the end of treatment and during the follow-up period, and analysed to determine how the risk of TB sequelae is linked with the socioeconomic position of the patient, to establish the occurrence of catastrophic costs due to TB and the proportion of patients that resort to potentially irreversible socioeconomic coping strategies.

Accurate data source will be maintained and confidentiality will be guaranteed. Data will be analysed according to the statistical plan. Results of the study will be disseminated to all relevant stakeholders through meetings, reports and publications.

ELIGIBILITY:
Inclusion Criteria:

* At least one sputum sample tested positive for Mtb by Xpert MTB/RIF assay in the study clinic/study laboratory or at least one sputum sample tested positive by culture methods in study laboratory or other TB laboratory
* Be ≥ 18 years of age
* Willingness to provide a written consent or witnessed oral consent in the case of illiteracy for participation in the study, prior to patient's first sample or other study-specific data being collected
* Willing to be tested for HIV infection
* Agrees to the collection and storage of blood, urine, and sputum specimens for use in future research
* Willing to start anti-TB treatment after TB diagnosis
* Living within the study area and willing to inform the study team of any change of address during the treatment and follow-up period

Exclusion Criteria:

* Has received TB treatment in the last 6 months
* Has incapacity to produce and provide two sputum samples of sufficient quality (3 ml)
* Has severe medical or psychiatric condition which in the opinion of the site investigator or designee, might interfere with the ability to give true informed consent and to adhere to the study requirements
* Is currently imprisoned
* Taking part in investigational product trials related to TB and/or lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a multi-country, multi-centre observational cohort study, conducted at four recruiting sites in four African countries: 1) University of the Witwatersrand (WITS), Johannesburg in South Africa; 2) NIMR-Mbeya Medical Research Center (NIMR-MMRC), Mbeya in Tanzania; 3) Instituto Nacional de Saúde (INS), Ministry of Health, Mozambique; 4) Medical Research Council (MRC) Unit The Gambia, Fajara, The Gambia.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe pulmonary function impairment | 2 years
  Measured by spirometry

SECONDARY OUTCOMES:
Changes in impairment of pulmonary function | 2 years
  Measured by six minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Gavin J Churchyard, Principal Investigator — Chief Executive Officers
Locations (4):
- Instituto Nacional de Saúde, Maputo, Mozambique
- The Clinical HIV Research Unit, Johannesburg, Gauteng, South Africa
- NIMR-Mbeya Medical Research Centre, Mbeya, Tanzania
- The MRC-Unit, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
To be shared amongst the Collaborators, on shared database when the study starts

REFERENCES:
- [Derived] Rachow A, Ivanova O, Wallis R, Charalambous S, Jani I, Bhatt N, Kampmann B, Sutherland J, Ntinginya NE, Evans D, Lonnroth K, Niemann S, Schaible UE, Geldmacher C, Sanne I, Hoelscher M, Churchyard G. TB sequel: incidence, pathogenesis and risk factors of long-term medical and social sequelae of pulmonary TB - a study protocol. BMC Pulm Med. 2019 Jan 7;19(1):4. doi: 10.1186/s12890-018-0777-3. PMID 30616617
- See also: TB Sequel Website — http://tbsequel.org